CLINICAL TRIAL: NCT07087717
Title: A Prospective Randomized Clinical Split-mouth Study on the Influence of Implant Surface Roughness on Peri-implant Bone Stability of Implants Supporting a Mandibular Overdenture.
Brief Title: Comparison of Implants With Different Implant Surfaces.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2014/1231/AM01 BC-8296
Record Dates: First submitted 2025-06-26; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Oral Health Quality of Life (OHQoL) Was Assessed; the Effect of Surface Roughness on Crestal Bone Remodelling; The Effect of Surface Roughness on Peri-implant Health
Keywords: implant surface; implant-supported overdenture; oral health quality of life; implant survival; hybrid implants; moderately rough implants

STUDY DESIGN:
Intervention Model Description: In this split-mouth randomized controlled trial patients received a mandibular overdenture supported by 2 different implants. One implant had a moderately rough surface (DCC) and one implant had a hybrid surface (MSC).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DCC-implant (Active Comparator): Implant with a moderatley rough surface (DCC) was placed in one part of the mandible.
  Interventions: Device: Split-Mouth Placement of an implant with a moderately rough surface (DCC).
- MSC-implant (Experimental): Implant with a a hybrid surface (MSC) was placed in a second part of the mandible.
  Interventions: Device: Split-Mouth Placement of an implant with a hybrid surface (MSC).

INTERVENTIONS:
Device: Split-Mouth Placement of an implant with a moderately rough surface (DCC). — Surgical placement of a dental implant in canine area (left or right, assigned by flipping a coin) of the mandibular bone of the patient.
  Arms: DCC-implant
Device: Split-Mouth Placement of an implant with a hybrid surface (MSC). — Surgical placement of a dental implant in canine area (left or right, assigned by flipping a coin) of the mandibular bone of the patient.
  Arms: MSC-implant

SUMMARY:
This study looks at how the surface texture of dental implants affects the surrounding bone and the overall gum health over time. It compares two types of implant surfaces: one partially smooth and one slightly rough. The researchers also check how these implant treatments impact patients' quality of life related to oral health after 1 year and again after 8 years.

DETAILED DESCRIPTION:
This split-mouth randomized controlled trial aimed to assess the effect of surface roughness on long-term crestal bone remodelling and peri-implant health, comparing hybrid and moderately rough implants. As a secondary aim, Oral Health Quality of Life (OHQoL) was assessed after 1 and 8 function years.

ELIGIBILITY:
Inclusion Criteria:

* Totally edentulous for at least four months
* Sufficient residual bone volume to place two implants of 4 mm in diameter and 9-11 mm in length

Exclusion Criteria:

* <21 years old
* Smoking
* General contra-indications for oral surgery, e.g., full-dose head and neck radiation, intravenously administrated bisphosphonates and current chemotherapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
The effect of surface roughness on long-term crestal bone remodelling. | From enrollment until 8 years.
  The effect of surface roughness on long-term crestal bone remodelling is evaluated by recording crestal bone loss (mm) on intra-oral periapical radiographs of the implants.

SECONDARY OUTCOMES:
Oral Health Quality of Life (OHQoL) | Assessed after 1 and 8 function years.
  The patients were asked to complete an Oral Health Impact Profile-14 (OHIP-14) questionnaire. Score varies beween min.0 and max.56. Lower values indicate better conditions.
Peri-implant Health: Probing pocket depth | At one year, 6 years, 8 years and 10 years of follow-up
  Probing pocket depth (mm) at 4 sites around the implant
Peri-implant health: Bleeding on probing | At one year, 6 years, 8 years and 10 years of follow-up.
  Bleeding on probing (yes/no) at 4 sites around the implant
Peri-implant Health: Plaque | at one year, 6 years, 8 years and 10 years of follow-up.
  Plaque (yes/no) at 4 sites around the implant

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Glibert, DDS, MSc, PhD, Principal Investigator — University Ghent
Locations (1):
- Oral Health Sciences - Department of Periodontology and Oral Implantology - P8, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glibert M, Matthys C, Maat RJ, De Bruyn H, Vervaeke S. A randomized controlled clinical trial assessing initial crestal bone remodeling of implants with a different surface roughness. Clin Implant Dent Relat Res. 2018 Oct;20(5):824-828. doi: 10.1111/cid.12652. Epub 2018 Jul 26. PMID 30048048